CLINICAL TRIAL: NCT00594672
Title: Age-Related Eye Disease Study (AREDS) and AREDS2 Follow-Up
Brief Title: Age-Related Eye Disease Study (AREDS) Follow-Up
Status: Active, not recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080043; 08-EI-0043
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-08-18

CONDITIONS: Age-Related Macular Degeneration; Cataract
Keywords: Cataract; Age-Related Macular Degeneration; Age-Related Macular Degeneration (AMD); Cataracts; Natural History; Age Related Macular Degeneration; AMD
MeSH Terms: conditions — Macular Degeneration; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AREDS participants: Participants who were enrolled in the AREDS or AREDS2 protocol and successfully completed the final AREDS or AREDS2 follow-up visit.

SUMMARY:
This study is a 5-year extension of the AREDS protocol, in which investigators followed the natural course of age-related macular degeneration (AMD) and cataracts. Participants in the former AREDS protocol are eligible for this study.

Participants have a complete eye examination once a year and are contacted at least once a year between visits to check on their status. The eye examination includes measurement of visual acuity (vision chart test) and examination of the inside of the eye after the pupils have been dilated with eye drops. Photographs of the inside of the eye may be taken using a special camera that flashes a bright light in the eye. A blood sample may be obtained to test for cholesterol level and genes related to inflammation.

DETAILED DESCRIPTION:
The Age-Related Eye Disease Study (AREDS) Follow-Up protocol allows us to continue with the follow-up of participants who were enrolled in the clinical trial of antioxidant vitamins and zinc. The AREDS study was designed in the beginning to determine the clinical course and prognosis of age-related macular degeneration (AMD) and cataracts.1 In addition, AREDS evaluated the possible risk factors associated with the development of AMD and cataracts; the nutritional risk factors were evaluated and published in October 2001.

Study results showed that antioxidant vitamins and zinc therapy reduced the risk of developing advanced AMD in participants with intermediate and greater risk of developing AMD (categories 3 and 4) by 25%. The risk of vision loss of three lines or more on the logarithmic visual acuity charts was also reduced by 19% for these participants. For those who developed AMD, their risk of vision loss was reduced by 25%. Antioxidants and zinc are now recommended for participants who have an intermediate risk of developing advanced AMD.

Upon completion of the AREDS clinical trial in September 2001, participants were invited for follow-up for an additional five years to collect further data on the natural course of both AMD and cataracts. Although the multi-center trial was complete in December 2005, we wish to continue to follow-up on these participants at the NEI on an annual basis for a minimum of five years from the date of enrollment in this study to collect additional data.

Although results from AREDS on the relationship of lutein/zeaxanthin and omega-3 long-chain polyunsaturated fatty acid (LCPUFA) intake with advanced AMD were informative, the non-experimental sampling (observational) design limited our strength of inference. AREDS2, a multi-center Phase III randomized clinical trial, was designed to assess the effects of oral supplementation of high doses of macular xanthophylls (lutein and zeaxanthin) and/or omega-3 LCPUFAs as a treatment for AMD, cataract, and moderate vision loss. In addition to this objective, the study provided information on the clinical course, prognosis, and risk factors for development and progression of both AMD and cataract. Other study goals included the evaluation of eliminating beta-carotene and/or reducing zinc in the original AREDS formulation on the progression and development of AMD. AREDS2 also sought to validate the fundus photographic AMD scale developed from AREDS. Participants who completed AREDS2 are invited for follow-up on an annual basis for at least five years from the date of enrollment in this study to collect additional data.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be eligible if they:

* Were enrolled in the AREDS or AREDS2 protocol and successfully completed the final AREDS or AREDS2 follow-up visit.
* Can understand and provide informed consent.

EXCLUSION CRITERIA:

Participants will not be eligible if they:

* Are under the age of 50.
* Are not able to return to NIH for examination for the duration of the trial.
* Have any systemic diseases that compromise the ability to provide adequate ophthalmologic examination.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who were enrolled in the AREDS or AREDS2 protocol and successfully completed the final AREDS or AREDS2 follow-up visit.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2008-06-02 (Actual)

PRIMARY OUTCOMES:
Outcomes assessed will be based on the ongoing ocular examination and historical data that will be obtained at each visit. The visual acuity data and the photographic documentation of the two diseases will be of particular importance. | 5 years
  Data on possible ocular events for both AMD and cataracts and for documentation of any adverse effects associated with the AREDS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seddon JM, De D, Rosner B. The role of nutritional factors in transitioning between early, mid, and late stages of age-related macular degeneration: prospective longitudinal analysis. Am J Clin Nutr. 2024 Dec;120(6):1387-1398. doi: 10.1016/j.ajcnut.2024.08.019. Epub 2024 Aug 23. PMID 39181206
- [Derived] Seddon JM, Silver RE, Rosner B. Response to AREDS supplements according to genetic factors: survival analysis approach using the eye as the unit of analysis. Br J Ophthalmol. 2016 Dec;100(12):1731-1737. doi: 10.1136/bjophthalmol-2016-308624. Epub 2016 Jul 28. PMID 27471039
- [Derived] Merle BM, Silver RE, Rosner B, Seddon JM. Dietary folate, B vitamins, genetic susceptibility and progression to advanced nonexudative age-related macular degeneration with geographic atrophy: a prospective cohort study. Am J Clin Nutr. 2016 Apr;103(4):1135-44. doi: 10.3945/ajcn.115.117606. PMID 26961928
- [Derived] Merle BM, Silver RE, Rosner B, Seddon JM. Adherence to a Mediterranean diet, genetic susceptibility, and progression to advanced macular degeneration: a prospective cohort study. Am J Clin Nutr. 2015 Nov;102(5):1196-206. doi: 10.3945/ajcn.115.111047. Epub 2015 Oct 21. PMID 26490493
- [Derived] Sangiovanni JP, Agron E, Meleth AD, Reed GF, Sperduto RD, Clemons TE, Chew EY; Age-Related Eye Disease Study Research Group. omega-3 Long-chain polyunsaturated fatty acid intake and 12-y incidence of neovascular age-related macular degeneration and central geographic atrophy: AREDS report 30, a prospective cohort study from the Age-Related Eye Disease Study. Am J Clin Nutr. 2009 Dec;90(6):1601-7. doi: 10.3945/ajcn.2009.27594. Epub 2009 Oct 7. PMID 19812176
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-EI-0043.html